CLINICAL TRIAL: NCT02694796
Title: Long Term Impact of a Physical Activity Intervention Combining Workshop During a Balneotherapy and a Web and Smartphone-based Physical Activity Program After Balneotherapy, on Physical Activity Level : a Randomized Control Trial
Brief Title: Impact of Web and Smartphone-based Physical Activity Program on Physical Activity Level 12 Months After a Balneotherapy
Acronym: THERMACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C2015/02
Record Dates: First submitted 2016-02-18; First posted 2016-03-01 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Physical Activity; Chronic Diseases; Obesity; Diabetes; Rheumatic Diseases; Cardiovascular Diseases; Breast Cancer; Chronic Obstructive Pulmonary Disease
Keywords: Web and smartphone-based physical activity program; Connected devices; Balneotherapy
MeSH Terms: conditions — Motor Activity; Chronic Disease; Obesity; Diabetes Mellitus; Rheumatic Diseases; Cardiovascular Diseases; Breast Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The 'Physical activity program after a balneotherapy' intervention involves providing a workshop during a balneotherapy about physical activity and use of automated physical activity program including website, mobile app and connected devices, and after the balneotherapy, the access to the automated program during 12 months.
  Interventions: Behavioral: Physical activity program after a balneotherapy
- Control (No Intervention): Patients included in the control arm will receive a booklet including informations about physical activity recommendations and practice.

INTERVENTIONS:
Behavioral: Physical activity program after a balneotherapy — workshop during the balneotherapy associated to an automated program of physical activity after the end of the balneotherapy available during 12 months
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the impact of an intervention combining a workshop during a balneotherapy and the use after the end of the balneotherapy of a web and smartphone-based physical activity program using connected devices, on physical activity level among patients 12 months after they participated in a balneotherapy in thermal care center.

A multi center randomized controlled trial is setting to evaluate the impact of the intervention on physical activity recommendations achievement of the patients.

Investigators hypothesize that an intervention including a workshop during a balneotherapy and an automated physical activity program using web, mobile phone and connected devices will help patients to be engaged in more physical activities and to reach physical activity recommendations.

DETAILED DESCRIPTION:
New technologies such as mobile phone and connected devices have been recognized as useful tools to assist chronic patients in their disease's management. they are also considering as promising tools to help patients to change their lifestyle behavior.

Balneotherapy is a very special moment to initiate changes and to raise awareness about healthier behavior in terms of food and physical activity.

The objective of the intervention is to help patients with chronic diseases, taking part in a balneotherapy, to increase or maintain their physical activity level in the long term to reach the national recommendations of 150 minutes of moderate physical activity per week.

Patients will be randomized either in the intervention group or in the control group.

The intervention group will participate in a workshop during the balneotherapy providing them informations about physical activity and also about the way to use the web and smartphone-based physical activity program along with the use of the connected devices (scale and pedometer). After the end of the balneotherapy, the intervention group will have access to the web and smartphone-based physical activity program during 12 months.

The control group will receive a booklet including informations about physical activity practice.

ELIGIBILITY:
Inclusion Criteria:

* age between 50 and 79
* BMI between 19 and 35 kg.m2
* stabilized chronic disease : cardiovascular disease, obesity, diabetes, chronic obstructive pulmonary disease, rheumatic diseases, breast cancer
* practice of moderate physical activity less than 150 minutes per week
* practice of sportive activity less than 2h per week
* having access to internet
* possessing a smartphone connected to internet
* good comprehension of french
* notice and informed consent signed
* no contraindication to practice physical activity
* subject to French Social Security

Exclusion Criteria:

* wearing a cardiac pacemaker
* non-stabilized chronic disease
* invalidating pathology of locomotor system
* metastatic cancers
* being in an exclusion period for participating in another study or having received more than 4500€ during the year due to participation in clinical studies
* being under supervision
* refusing to be register in the French National Volunteers Register

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Achievement of Physical activity recommendations | at 12 months of follow-up
  Proportion of patients in each arm of the study (intervention and control) who achieve physical activity recommendations.
  Physical activity will be measured by IPAQ questionnaire (International Physical Activity Questionnaire). Achievement of physical activity recommendations corresponds to 150 minutes of moderate physical activity per week.
  To compare physical activity at 12 months, a constrained Longitudinal Data Analysis will be used involving the repeated measure of physical activity at inclusion and every 2 months until the end of the 12 months of follow-up.

SECONDARY OUTCOMES:
Physical activity | at inclusion, 6 and 12 months of follow-up
  IPAQ questionnaire to evaluate in each arm of the study physical activity (like physical activity level, sedentary time, the proportion of patients reporting an increase of at least 20 minutes of moderate physical activity per week)
Weight | at inclusion, 6 and 12 months of follow-up
Waist circumference | at inclusion, 6 and 12 months of follow-up
Quality of life | at inclusion, 6 and 12 months of follow-up
  The quality of life will be measured thanks to the SF-12 questionnaire (Short Form Health Survey)
Captured physical activity | at return home after the end of the balneotherapy, at 6 months and at 12 months of follow-up
  Physical activity will be measured thanks to accelerometers integrated into smartphones

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire Gabriel Montpied, Clermont Ferrand
Locations (9):
- France (9):
  - Thermes CHEVALLEY, Aix-les-Bains
  - Centre thermal d'Amélie-les-Bains, Amélie-les-Bains
  - Thermes de Bourbon-Lancy, Bourbon-Lancy
  - Thermes de Brides-les-Bains, Brides-les-Bains
  - Caleden Complexe Thermal, Chaudes-Aigues
  - Centre thermal d'Eugénie-les-Bains, Eugénie-les-Bains
  - Thermes du Boulou, Le Boulou
  - Thermes de Vals-les-Bains, Vals-les-Bains
  - Thermes CALLOU, Vichy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Weegen S, Verwey R, Spreeuwenberg M, Tange H, van der Weijden T, de Witte L. It's LiFe! Mobile and Web-Based Monitoring and Feedback Tool Embedded in Primary Care Increases Physical Activity: A Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Jul 24;17(7):e184. doi: 10.2196/jmir.4579. PMID 26209025
- [Background] Aalbers T, Baars MA, Rikkert MG. Characteristics of effective Internet-mediated interventions to change lifestyle in people aged 50 and older: a systematic review. Ageing Res Rev. 2011 Sep;10(4):487-97. doi: 10.1016/j.arr.2011.05.001. Epub 2011 May 20. PMID 21628005
- [Background] Ammann R, Vandelanotte C, de Vries H, Mummery WK. Can a website-delivered computer-tailored physical activity intervention be acceptable, usable, and effective for older people? Health Educ Behav. 2013 Apr;40(2):160-70. doi: 10.1177/1090198112461791. Epub 2012 Oct 16. PMID 23077157
- [Background] Martin SS, Feldman DI, Blumenthal RS, Jones SR, Post WS, McKibben RA, Michos ED, Ndumele CE, Ratchford EV, Coresh J, Blaha MJ. mActive: A Randomized Clinical Trial of an Automated mHealth Intervention for Physical Activity Promotion. J Am Heart Assoc. 2015 Nov 9;4(11):e002239. doi: 10.1161/JAHA.115.002239. PMID 26553211
- [Background] Krebs P, Prochaska JO, Rossi JS. A meta-analysis of computer-tailored interventions for health behavior change. Prev Med. 2010 Sep-Oct;51(3-4):214-21. doi: 10.1016/j.ypmed.2010.06.004. Epub 2010 Jun 15. PMID 20558196
- [Background] Irvine AB, Gelatt VA, Seeley JR, Macfarlane P, Gau JM. Web-based intervention to promote physical activity by sedentary older adults: randomized controlled trial. J Med Internet Res. 2013 Feb 5;15(2):e19. doi: 10.2196/jmir.2158. PMID 23470322
- [Derived] Fillol F, Paris L, Pascal S, Mulliez A, Roques CF, Rousset S, Duclos M. Possible Impact of a 12-Month Web- and Smartphone-Based Program to Improve Long-term Physical Activity in Patients Attending Spa Therapy: Randomized Controlled Trial. J Med Internet Res. 2022 Jun 16;24(6):e29640. doi: 10.2196/29640. PMID 35708743